CLINICAL TRIAL: NCT01940081
Title: The Leiden Nonischemic Cardiomyopathy Study
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Katja Zeppenfeld, Prof. dr., Leiden University Medical Center
Other Study IDs: Cardiomyopathy study
Record Dates: First submitted 2013-08-29; First posted 2013-09-11 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Cardiomyopathy, Dilated; Tachycardia, Ventricular; Ventricular Fibrillation
Keywords: Cardiomyopathy, Dilated; Tachycardia, Ventricular; Ventricular Fibrillation; Arrhythmias, Cardiac/etiology; Arrhythmias, Cardiac/physiopathology; Magnetic Resonance Imaging; 3-Iodobenzylguanidine/diagnostic use; Sympathetic Nervous System/radionuclide imaging; Electrophysiologic Techniques, Cardiac; Biopsy; Genetic Testing; Echocardiography; Electrocardiography, Ambulatory; Exercise Test
MeSH Terms: conditions — Cardiomyopathy, Dilated; Tachycardia, Ventricular; Ventricular Fibrillation; Arrhythmias, Cardiac | interventions — Exercise Test; Blood Specimen Collection; Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Per patient:
  Blood samples (40 mL) Ventricular biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group A: Nonischemic cardiomyopathy - not admitted for surgery: Patients with nonischemic cardiomyopathy with:
  * documented ventricular arrhythmia or
  * suspected ventricular arrhythmia (e.g. because of out-of-hospital cardiac arrest, palpitations or syncope) or
  * high risk for ventricular arrhythmia (LVEF ≤ 35%) or
  * intermediate risk for ventricular arrhythmia (LVEF ≤ 50% and late enhancement on contrast-enhanced MRI)
  who are not admitted for cardiac surgery
  Interventions: Other: Transthoracic echocardiography; Other: Exercise test; Other: 24-hour Holter electrocardiogram; Other: Contrast-enhanced magnetic resonance imaging; Other: 123-iodine metaiodobenzylguanidine imaging; Other: Blood samples; Genetic: Genetic analysis; Procedure: Invasive electrophysiological study; Procedure: Endomyocardial biopsy
- Group B: Nonischemic cardiomyopathy -admitted for surgery: Patients with nonischemic cardiomyopathy with:
  * documented ventricular arrhythmia or
  * suspected ventricular arrhythmia (e.g. because of out-of-hospital cardiac arrest, palpitations or syncope) or
  * high risk for ventricular arrhythmia (LVEF ≤ 35%)
  who are admitted for cardiac surgery (e.g., mitral valve annuloplasty or CorCap)
  Interventions: Other: Transthoracic echocardiography; Other: Exercise test; Other: 24-hour Holter electrocardiogram; Other: Contrast-enhanced magnetic resonance imaging; Other: 123-iodine metaiodobenzylguanidine imaging; Other: Blood samples; Genetic: Genetic analysis; Procedure: Invasive electrophysiological study; Procedure: Intraoperative biopsy; Procedure: Intraoperative mapping and/or ablation
- Group C: Controls: Patients without nonischemic cardiomyopathy (controls) who are admitted for:
  * Coronary artery bypass graft surgery and who do not have prior myocardial infarction
  * Aortic valve replacement
  Interventions: Other: Transthoracic echocardiography; Other: Exercise test; Other: 24-hour Holter electrocardiogram; Other: Contrast-enhanced magnetic resonance imaging; Other: Blood samples; Procedure: Intraoperative biopsy

INTERVENTIONS:
Other: Transthoracic echocardiography
Other: Exercise test
Other: 24-hour Holter electrocardiogram
Other: Contrast-enhanced magnetic resonance imaging
Other: 123-iodine metaiodobenzylguanidine imaging
  Groups: Group A: Nonischemic cardiomyopathy - not admitted for surgery; Group B: Nonischemic cardiomyopathy -admitted for surgery
Other: Blood samples
Genetic: Genetic analysis
  Groups: Group A: Nonischemic cardiomyopathy - not admitted for surgery; Group B: Nonischemic cardiomyopathy -admitted for surgery
Procedure: Invasive electrophysiological study
  Groups: Group A: Nonischemic cardiomyopathy - not admitted for surgery; Group B: Nonischemic cardiomyopathy -admitted for surgery
Procedure: Endomyocardial biopsy
  Groups: Group A: Nonischemic cardiomyopathy - not admitted for surgery
Procedure: Intraoperative biopsy
  Groups: Group B: Nonischemic cardiomyopathy -admitted for surgery; Group C: Controls
Procedure: Intraoperative mapping and/or ablation
  Groups: Group B: Nonischemic cardiomyopathy -admitted for surgery

SUMMARY:
Rationale: Sudden cardiac death, mainly caused by ventricular arrhythmias (VA), is a major cause of morbidity and mortality in non-ischemic cardiomyopathy (NICM). Therapies that effectively prevent VA are lacking. Improved understanding of the substrate and mechanisms of VA in NICM may allow more effective, individualized and substrate-based therapies to be developed. In addition, risk stratification in NICM needs to be improved so that therapies can be allocated more efficiently.

Objectives: 1) To improve our understanding of the underlying pro-arrhythmic substrate and electrophysiologic mechanisms of VA in NICM, and to develop individualized treatment for VA based on the identified substrate. 2) To improve risk stratification for VA and sudden cardiac death in NICM based on substrate characteristics. 3) to evaluate disease progression in NICM.

Hypothesis: Improved understanding of the substrate and mechanisms of VA in NICM may allow more effective, individualized and substrate-based therapies to be developed.

Study design: A prospective cohort study.

Study population: The study population will consist of three groups (A, B and C): NICM patients with documented VA, suspected VA or intermediate to high risk for VA (according to established criteria) who are not referred for cardiac surgery (group A), NICM patients with documented VA, suspected VA or a high risk for VA who are referred for cardiac surgery (group B) and a control group consisting of patients without NICM who are referred for cardiac surgery (group C).

Evaluation: All patients will be evaluated according to current standards for patients with NICM. Evaluation will include 24h-Holter, echocardiography, coronary angiogram and contrast-enhanced MRI (CE-MRI). If CE-MRI is performed in another hospital, additional recordings will be performed in our hospital. Additionally, blood samples (arterial, cardiac venous and peripheral venous) for collagen turnover markers will be taken from all patients. 123-iodine metaiodobenzylguanidine (123-I MIBG) imaging, electrophysiologic study and endomyocardial biopsy will be performed in group A and B. Intra-operative biopsy will be performed in group B and C.

Intervention: In group B, intra-operative mapping and cryo-ablation and postoperative electrophysiologic study will be performed in patients with subepicardial late enhancement on MRI or induced VA suspected for an subepicardial origin.

Main study parameters/endpoints: The main study parameters are extent, location and pattern of fibrosis on imaging and in biopsy specimens. The main study endpoints are inducibility of VA, type of induced VA, spontaneous VA and type of spontaneous VA.

ELIGIBILITY:
Inclusion criteria, group A:

* Nonischemic cardiomyopathy
* Documented ventricular arrhythmia, suspected ventricular arrhythmia (e.g. because of out-of-hospital cardiac arrest, palpitations or syncope) or high risk for ventricular arrhythmias (LVEF ≤ 35%) or intermediate risk for ventricular arrhythmias (LVEF ≤ 50% and late enhancement on contrast-enhanced MRI)
* Admission not for cardiac surgery

Inclusion criteria, group B:

* Nonischemic cardiomyopathy
* Documented ventricular arrhythmia or suspected ventricular arrhythmia (e.g. because of out-of-hospital cardiac arrest, palpitations or syncope) or high risk for ventricular arrhythmia (LVEF ≤ 35%)
* Admission for cardiac surgery (e.g., mitral valve annuloplasty or CorCap)

Inclusion criteria, group C:

- Patients undergoing aortic valve replacement or coronary artery bypass graft surgery

Exclusion criteria, all groups:

* Age < 18 years or > 80 years
* Inadequate patient competence
* Pregnancy
* Inability to comply with the protocol due to haemodynamic instability

Exclusion Criteria, groups A and B:

- Other cardiomyopathy (e.g., prior myocardial infarction, infiltrative cardiac disease such as sarcoidosis, amyloidosis or Chagas cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy/dysplasia, hypertrophic cardiomyopathy, non-compaction cardiomyopathy and congenital heart disease)

Exclusion criteria, group C:

* Nonischemic cardiomyopathy
* Prior myocardial infarction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with nonischemic cardiomyopathy and controls who are admitted to the hospital
Sampling Method: Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Inducibility of ventricular arrhythmias | Baseline electrophysiological study
Type of induced ventricular arrhythmias | Baseline electrophysiological study
Spontaneous ventricular arrhythmias | Up to 10 years
Type of spontaneous ventricular arrhythmias | Up to 10 years

SECONDARY OUTCOMES:
Hospital admissions for heart failure | Up to 10 years
Cardiac mortality | Up to 10 years
All-cause mortality | Up to 10 years
LV function/dimensions/compact fibrosis deterioration as assessed by 123-I MIBG imaging and/or CE-MRI | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Cardiology, Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Derived] Piers SR, Androulakis AF, Yim KS, van Rein N, Venlet J, Kapel GF, Siebelink HM, Lamb HJ, Cannegieter SC, Man SC, Zeppenfeld K. Nonsustained Ventricular Tachycardia Is Independently Associated With Sustained Ventricular Arrhythmias in Nonischemic Dilated Cardiomyopathy. Circ Arrhythm Electrophysiol. 2022 Feb;15(2):e009979. doi: 10.1161/CIRCEP.121.009979. Epub 2022 Jan 28. PMID 35089806